CLINICAL TRIAL: NCT00621062
Title: Randomized Prospective Trial of Varicose Vein Surgery
Brief Title: Prospective Randomized Trial Comparing the New Endovenous Procedures Versus Conventional Surgery for Varicose Veins Due to Great Saphenous Vein Incompetence
Acronym: RAFPELS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Centrallasarettet Västerås (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RAFPELS
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2011-03

CONDITIONS: Varicose Veins
Keywords: varicose; vein; ligation; laser; foam; sclerotherapy; radiofrequency; duplex; sf36; Aberdeen; VCSS; quality; recurrence
MeSH Terms: conditions — Varicose Veins; Recurrence | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High Ligation of the GSV (Active Comparator)
  Interventions: Procedure: High Ligation of the GSV
- Endovenous Laser Ablation (Active Comparator)
  Interventions: Procedure: Endovenous Laser Ablation
- Radiofrequency ablation (Active Comparator)
  Interventions: Procedure: Radiofrequency ablation
- Foam Sclerotherapy (Active Comparator)
  Interventions: Procedure: Foam Sclerotherapy

INTERVENTIONS:
Procedure: High Ligation of the GSV — Performed in local or general anesthesia in accordance to clinical praxis and the patients own preference. After high ligation the GSV is stripped from the groin to the most distant insufficient part or just under the knee joint.All proximal branches are ligated. Including the superficial epigastric vein. The stripping instrument can be inserted in either cranial or caudal direction but all veins are stripped in the cranio-caudal direction.
  Arms: High Ligation of the GSV
Procedure: Endovenous Laser Ablation — Laser ablation is performed in tumescence anesthesia which is performed with a 150-200 ml (sometimes more is required, up to 400ml in patients with a poorly formed saphenous sheath) solution of lidocaine with adrenaline supplement. General sedation can be administrated as a supplement (with intravenous Propofol or Dormicum when needed). Laser is performed under duplex guidance and the catheter is inserted percutaneously into the GSV at knee level and parked distant to the saphenofemoral junction (SFJ) just distal to the superficial epigastric vein. Laser ablation is performed down to the most distal insufficient part of GSV or just below the knee joint. We use an effect of 14 Watt administration of 70-80 J / cm at a continuous mode at a speed of 1cm/5sec.
  Arms: Endovenous Laser Ablation
Procedure: Radiofrequency ablation — RF ablation is performed in tumescence anesthesia which is performed with a 150-200 ml solution (same as above) of lidocaine with adrenaline supplement. General sedation can be administrated as a supplement (with intravenous Propofol or Dormicum when needed). RF is performed under duplex guidance and the Closure-FAST catheter is inserted percutaneously into the GSV at the knee level and parked distant to the SFJ just distal to the superficial epigastric vein. Probe size and length used for RF is chosen in accordance to the manufacturer's recommendation and with a probe temperature of 120 degrees C. RF closure is performed down to the most distal insufficient part of GSV or just under the knee joint.
  Arms: Radiofrequency ablation
Procedure: Foam Sclerotherapy — Sclerosant foam consists of 2ml 3% aethoxysclerol mixed with 8ml air (Tessari method). A maximum of 10 ml is injected. Access to the vein for the sclerosant is gained by a duplex guided puncture or a mini incision mid-thigh or just above the knee and the amount of sclerosant foam used is 2,5-10 ml. Duplex is used prior to the operation in order to mark the vein and during the operation in order to control the extent of the sclerofoam. Duplex validates that foam is deposed to the whole length of the GSV. Blood from the veins is drained by means of elevation prior to the deposition of the sclerofoam. The leg is then bandaged with elastic bandage.
  Arms: Foam Sclerotherapy

SUMMARY:
Through a prospective RCT evaluate and compare the three new endovenous methods for great saphenous vein ablation (Radiofrequency, endovenous laser and foam sclerotherapy) versus high ligation and stripping. Procedure (proof-of-concept) and patient related (clinical outcome) factors will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Clinical examinations by an experienced surgeon as well as duplex evaluation. Duplex evaluation of both the deep and the superficial system is required but not of the perforating vessels. It is performed by experienced BMA or surgeon with profound knowledge in vein diagnosis with duplex.
* Patients with primary varicose vein disease between age 18 to 75.
* Signature of informed consent.
* Varicose veins and duplex verified GSV incompetence defined as >0,5 seconds reflux time after manual compression in upright position 60 degrees.
* Vein size <20 mm in upright position 60 degrees, 2 cm below the SFJ.
* Minimum distance between skin and the GSV in the first 20 cm from the SFJ > 5mm.
* CEAP classification C2-C5
* BMI <35

Exclusion Criteria:

* Non-consent for randomisation.
* Age <18 years.
* Age >75 years.
* Deep vein insufficiency in the same extremity (duplex verified).
* Vein size >20mm in upright position 60 degrees below the SFJ.
* Meander and superficial veins with a distance of <5mm to the skin surface ( RF or Laser cannot be applied).
* Patients with double GSV's and/or lateral accessory insufficient branch.
* Patients with cognitive disturbances, dementia or unable to understand for any reason the importance of follow up.
* Earlier operation with HL/S (recurrency).
* Operated for small saphenous vein (SSV) incompetence the last 3 months.
* Known ABI <0,9 or history of intermittent claudication or peripheral pulselessness (clinical examination)in either extremity.
* Patients with recent cancer diagnosis or undergoing cancer treatment.
* BMI >35.
* Patients with other known medical condition that contradict any of the treatments in the study.
* Minimum distance between skin and the GSV in the first 20 cm from the SFJ >5mm.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2008-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Recurrence rate and complications after venous surgery. Duplex ultrasound and clinical evaluation. | 3 years

SECONDARY OUTCOMES:
Quality of Life with SF36, Aberdeen Vein Score, VCSS and Visual Analogue Scale Scoring. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anders Hellberg, MD, PhD, Principal Investigator — Dept. of Vascular Surgery, Central Hospital of Västerås; Adam Bersztel, MD, PhD, Principal Investigator — Dept. of Vascular Surgery, Central Hospital of Västerås; Jerszy Leppert, Professor, Study Chair — Västerås Centrum for Clinical Research, University of Uppsala; Achilleas Karkamanis, MD, Principal Investigator — Dept. of Vascular Surgery, Central Hospital of Västerås
Locations (1):
- Department of Vascular Surgery; Central Hospital of Västerås, Västerås, Sweden